CLINICAL TRIAL: NCT01147224
Title: Alvesco for the Therapy of Persistent Asthma With or Without Allergic Component
Brief Title: ATEM (Alvesco Non-interventional Study)
Acronym: ATEM
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-9709-401-DE
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-09

CONDITIONS: Asthma; Allergy
Keywords: Asthma; Allergy; Ciclesonide; Alvesco; Inhaled steroids
MeSH Terms: conditions — Asthma; Hypersensitivity | interventions — ciclesonide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ATEM: A prospective one-arm non-interventional study with asthma patients treated with Alvesco.
  Interventions: Drug: Alvesco

INTERVENTIONS:
Drug: Alvesco — This is an observational study. Therefore, the physician decides about dosage according to individual needs.
  Other Names: Ciclesonide

SUMMARY:
The aim of the study is to evaluate the efficacy of Alvesco in patients with persistent asthma including or excluding allergic components over 3 months, especially in the spring season. Alvesco will be inhaled by a metered-dose inhaler. The study will provide further data on safety and tolerability of Alvesco .

ELIGIBILITY:
Main Inclusion Criteria:

* Asthma with or without allergic components

Main Exclusion Criteria:

* Hypersensitive to compounds of Alvesco
* Other criteria as defined in the Summary of Product Characteristics, Chapter 4.3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Treatment success with Alvesco | after 3 months
  Pre-/ post comparison of FEV1, Quality of life, Patient Questionnaire

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (66):
- Austria (66):
  - Nycomed Pharma GmbH, Amstetten
  - Nycomed Pharma GmbH, Baden
  - Nycomed Pharma GmbH, Bludenz
  - Nycomed Pharma GmbH, Böhlerwerk
  - Nycomed Pharma GmbH, Braunau am Inn
  - Nycomed Pharma GmbH, Bregenz
  - Nycomed Pharma GmbH, Dornbirn
  - Nycomed Pharma GmbH, Enns
  - Nycomed Pharma GmbH, Feldbach
  - Nycomed Pharma GmbH, Feldkirch
  - Nycomed Pharma GmbH, Furth
  - Nycomed Pharma GmbH, Gföhl
  - Nycomed Pharma GmbH, Gr. Siegharts
  - Nycomed Pharma GmbH, Graz
  - Nycomed Pharma GmbH, Graz-Gösting
  - Nycomed Pharma GmbH, Groß-Gerungs
  - Nycomed Pharma GmbH, Gunskirchen
  - Nycomed Pharma GmbH, Güssing
  - Nycomed Pharma GmbH, Haag
  - Nycomed Pharma GmbH, Hall in Tirol
  - Nycomed Pharma GmbH, Hallein
  - Nycomed Pharma GmbH, Hartberg
  - Nycomed Pharma GmbH, Herzogenburg
  - Nycomed Pharma GmbH, Innsbruck
  - Nycomed Pharma GmbH, Judenburg
  - Nycomed Pharma GmbH, Kaltenbach
  - Nycomed Pharma GmbH, Kirchdorf and Der Krems
  - Nycomed Pharma GmbH, Kitzbühel
  - Nycomed Pharma GmbH, Klein-Pöchlam
  - Nycomed Pharma GmbH, Landeck
  - Nycomed Pharma GmbH, Leibnitz, Styria
  - Nycomed Pharma GmbH, Lenzing
  - Nycomed Pharma GmbH, Linz
  - Nycomed Pharma GmbH, Litschau
  - Nycomed Pharma GmbH, Mank
  - Nycomed Pharma GmbH, Melk
  - Nycomed Pharma GmbH, Mittersill
  - Nycomed Pharma GmbH, Mödling
  - Nycomed Pharma GmbH, Mühldorf
  - Nycomed Pharma GmbH, Münster
  - Nycomed Pharma GmbH, Neumarkt am Wallersee
  - Nycomed Pharma GmbH, Niederkreuzstetten
  - Nycomed Pharma GmbH, Pasching
  - Nycomed Pharma GmbH, Pinkafeld
  - Nycomed Pharma GmbH, Pucking
  - Nycomed Pharma GmbH, Saint Johann I. Pg.
  - Nycomed Pharma GmbH, Salzburg
  - Nycomed Pharma GmbH, Sankt Pölten
  - Nycomed Pharma GmbH, Schlüsslberg
  - Nycomed Pharma GmbH, Schörfling
  - Nycomed Pharma GmbH, Schwanenstadt
  - Nycomed Pharma GmbH, St.Georgen i.A.
  - Nycomed Pharma GmbH, Steyr
  - Nycomed Pharma GmbH, Strallegg
  - Nycomed Pharma GmbH, Sulz
  - Nycomed Pharma GmbH, Thalheim bei Wels
  - Nycomed Pharma GmbH, Traisen
  - Nycomed Pharma GmbH, Traismauer
  - Nycomed Pharma GmbH, Vienna
  - Nycomed Pharma GmbH, Voitsberg
  - Nycomed Pharma GmbH, Waidhofen/Thaya
  - Nycomed Pharma GmbH, Weitra
  - Nycomed Pharma GmbH, Wiener Neustadt
  - Nycomed Pharma GmbH, Wilhelmsburg
  - Nycomed Pharma GmbH, Ysper
  - Nycomed Pharma GmbH, Zwettl Stadt